CLINICAL TRIAL: NCT00561717
Title: A Four-Way Double-Blind, Randomized, Placebo Controlled Study to Determine the Efficacy and Speed of Azelastine Nasal Spray and Antihistaminic Agents in Adult Subjects With Allergen Induced Seasonal Allergic Rhinitis
Brief Title: A Randomized, Placebo Controlled Study to Determine the Efficacy and Speed of a Nasal Spray in Allergen Induced Seasonal Allergic Rhinitis
Acronym: GEYSER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Kingston Health Sciences Centre (Other)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Consumer Care Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 12962; 9427-B2171-22C (CR Number) (Other: company internal)
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Seasonal Allergic Rhinitis; Ragweed; Pollen; Allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity | interventions — azelastine; Loratadine; Cetirizine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Azelastine and placebo
- Arm 2 (Active Comparator)
  Interventions: Drug: Loratadine and Placebo
- Arm 3 (Active Comparator)
  Interventions: Drug: Cetirizine and Placebo
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo and Placebo (spray and Tablet)

INTERVENTIONS:
Drug: Azelastine and placebo — One Astelin spray per nostril plus one placebo tablet. In Cross-Over-Design with other arms.
  Arms: Arm 1
Drug: Loratadine and Placebo — One placebo spray per nostril plus one Loratadine 10 mg tablet. In Cross-Over-Design with other arms.
  Arms: Arm 2
Drug: Cetirizine and Placebo — One placebo spray per nostril plus one 10 mg Cetirizine tablet. In Cross-Over-Design with other arms.
  Arms: Arm 3
Drug: Placebo and Placebo (spray and Tablet) — One placebo spray per nostril plus one placebo tablet. In Cross-Over-Design with other arms.
  Arms: Arm 4

SUMMARY:
Finding out how fast azelastine nasal spray works in subjects with hay fever.

ELIGIBILITY:
Inclusion Criteria:

* History of seasonal allergic rhinitis to ragweed pollen for last 2 consecutive seasons;
* Positive response to skin prick test to ragweed allergen at screening;
* Be willing to participate in the trial.

Exclusion Criteria:

* History of hypersensitivity to azelastine;
* Females who are pregnant or lactating;
* Relative chronic sinusitis or nasal structural abnormalities causing greater than 50% obstruction;
* Asthma that requires other than occasional use of inhaled short-acting beta-2 antagonist;
* Known non-responsiveness to antihistamines;
* Alcoholism or drug abuse within 2 yrs. of screening;
* Current or regular use within 6 months of any type of tobacco product;
* Evidence of any clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic or malignancies within the last 5 years;
* History of a positive test to HIV, TB, hepatitis B or C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Onset of action measured by change in total nasal symptom score Until "Onset of action" = until drug demonstrates and maintains a change greater than placebo compared to baseline | Up to 6 hours

SECONDARY OUTCOMES:
Change from baseline for individual symptoms of allergic seasonal rhinitis; overall assessment of efficacy | Effect over 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kingston, Ontario, Canada

REFERENCES:
- [Derived] Tenn MW, Steacy LM, Ng CC, Ellis AK. Onset of action for loratadine tablets for the symptomatic control of seasonal allergic rhinitis in adults challenged with ragweed pollen in the Environmental Exposure Unit: a post hoc analysis of total symptom score. Allergy Asthma Clin Immunol. 2018 Jan 16;14:5. doi: 10.1186/s13223-017-0227-4. eCollection 2018. PMID 29371864